CLINICAL TRIAL: NCT03952507
Title: A Phase 1 Open-label Study in Healthy Subjects to Assess the Relative Oral Bioavailability and Food Effect of Single-dose JNJ-64417184 Administered as Tablets and as Suspension
Brief Title: A Study to Assess the Relative Oral Bioavailability and Food Effect of Single-dose of JNJ-64417184 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR108632; 64417184RSV1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 milligram (mg) oral tablet under fasted conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg oral tablet in fed conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg as oral suspension in fasted condition on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)
- Group 2: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 mg oral tablet under fed conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg as oral suspension in fasted conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg tablet under fasted conditions on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)
- Group 3: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 mg as oral suspension in fasted conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg tablet under fasted conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg tablet under fed conditions on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)
- Group 4: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 mg tablet under fasted conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg as oral suspension in fasted conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg tablet under fed conditions on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)
- Group 5: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 mg tablet under fed conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg tablet under fasted conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg as oral suspension in fasted conditions on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)
- Group 6: JNJ-64417184 (Experimental): Participants will receive JNJ-64417184 600 mg as oral suspension in fasted conditions on Day 1 in Treatment Period 1; followed by JNJ-64417184 600 mg tablet under fed conditions on Day 8 in Treatment Period 2; followed by JNJ-64417184 600 mg tablet under fasted conditions on Day 15 in Treatment Period 3. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184 600 (Oral Tablet Formulation); Drug: JNJ-64417184 (Oral Suspension Formulation)

INTERVENTIONS:
Drug: JNJ-64417184 600 (Oral Tablet Formulation) — Participants will receive 600 mg of JNJ-64417184 as oral tablet.
Drug: JNJ-64417184 (Oral Suspension Formulation) — Participants will also receive JNJ-64417184 600 mg as oral suspension.

SUMMARY:
The main purpose of this study is to evaluate the relative bioavailability of JNJ-64417184, formulated as a test formulation (tablet) compared to a reference formulation (suspension), administered orally in a fasted state, in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical and surgical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the hematology, biochemistry, blood coagulation, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must have a normal 12-lead electrocardiogram (ECG) (triplicate) at screening, including: normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate (QTc) according to Fridericia (QTcF) less than or equal to (<=) 450 milli second (ms) for male participants and <=470 ms for female participants; QRS interval less than (<) 120 ms; PR interval <=200 ms. If the results of the ECG are outside the normal ranges, the participant may be included only if the investigator judges the deviations from normal ECG to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Female participant must have a negative highly sensitive serum beta human chorionic gonadotropin (beta hCG) pregnancy test at screening and on Days -1, 7, and 14 (except for postmenopausal female participants)
* Female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after the last study drug intake

Exclusion Criteria:

* Past history of cardiac arrhythmias (example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Current human immunodeficiency virus (HIV)-type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A, B, or C infection, or current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen), or hepatitis C virus (HCV) infection (confirmed by HCV antibody) at screening
* A history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Known allergies, hypersensitivity, or intolerance to JNJ-64417184 or any of its excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2019-06-22 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability of JNJ-64417184 | Day 1,8,15:Predose, 0.5,1,2,3,4,6,8,10,12 and 18 hours (hrs) postdose; Day 2,9,16:24,36hrs postdose; Day 3,10,17:48 hrs postdose; Day 4,11,18:72hrs postdose; Day 5,12,19:96hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  The relative bioavailability based on Cmax, AUC(0last), and AUC(0-infinity) will be estimated as 100*Test/Reference where Test is tablet formulation of JNJ-64417184 and Reference is suspension formulation of JNJ-64417184 administered orally in a fasted state.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-64417184 in Fasted Conditions | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  Plasma concentration of JNJ-64417184 will be determined when administered as suspension under fasted conditions.
Plasma Concentration of JNJ-64417184 in fed and Fasted Conditions | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  Plasma concentration of JNJ-64417184 will be determined when administered as tablet under fed and fasted conditions.
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-64417184 in fed State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  Cmax is defined as maximum observed plasma analyte concentration of JNJ-64417184 in fed state.
Area Under the Plasma Analyte Concentration- time Curve from time 0 to time of the last Quantifiable Concentration (AUC [0-last]) in fed State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  AUC (0-last) is defined as area under the plasma analyte concentration- time curve (AUC) from time 0 to time of the last quantifiable concentration of JNJ-64417184 in fed state.
Area Under the Plasma Analyte Concentration-time Curve From time 0 to Infinite time (AUC [0-infinity]) in fed State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  AUC (0-infinity) is defined as area under the plasma analyte concentration-time curve (AUC) from time 0 to infinite time of JNJ-64417184 in fed state.
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-64417184 in Fasted State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  Cmax is defined as maximum observed plasma analyte concentration of JNJ-64417184 in fasted state.
Area Under the Plasma Analyte Concentration- time Curve from time 0 to time of the last (AUC [0-last]) Quantifiable Concentration in Fasted State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  AUC (0-last) is defined as area under the plasma analyte concentration- time curve (AUC) from time 0 to time of the last quantifiable concentration of JNJ-64417184 in fasted state.
Area Under the Plasma Analyte Concentration-time Curve From time 0 to Infinite time (AUC [0-infinity]) in Fasted State | Day 1,8,15:Predose, 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, and 18 hrs postdose; Day 2, 9, 16: 24, 36 hrs postdose; Day 3, 10, 17: 48 hrs postdose; Day 4, 11, 18: 72hrs postdose; Day 5, 12, 19: 96 hrs postdose;Day 6, 13, 20: 120hrs postdose up to Day 21
  AUC (0-infinity) is defined as area under the plasma analyte concentration-time curve (AUC) from time 0 to infinite time of JNJ-64417184 in fasted state.
Number of Participants with Adverse Event as Measure of Safety and Tolerability | Approximately 21 Days
  An adverse event is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Salt Lake City Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency